CLINICAL TRIAL: NCT00592995
Title: Creatine Safety and Tolerability in Premanifest HD: PRECREST
Acronym: PRECREST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven M. Hersch, Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006P001640; P01NS058793 (NIH)
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: Creatine monohydrate

INTERVENTIONS:
Drug: Creatine monohydrate — 10 to 30 grams daily
  Arms: 2
Drug: Placebo — 10 to 30 grams daily
  Arms: 1

SUMMARY:
PRECREST is a two phase protocol for Huntington's disease in which 60 premanifest and at-risk subjects will first be randomized into a double blind placebo controlled dose titration study bringing them to 30 grams daily or their highest tolerated dose. This phase will establish the highest tolerable doses in premanifest HD and permit the detection of toxicity and intolerability with attribution to active compound versus placebo, and enable a dose response assessment of biomarkers. In the second phase, all subjects will enter a year long open-label treatment on 30 grams daily (or their highest dose) of creatine to assess long term exposure to high dose creatine and its long term impact on various biomarkers.

DETAILED DESCRIPTION:
Extensive evidence exists that neurodegeneration begins many years before HD can be diagnosed clinically. Therefore, it is most desirable to begin a neuroprotective therapy before or during this premanifest period with the aim of delaying onset, as well as slowing functional decline. Cellular energy depletion is present early in HD and can be ameliorated by creatine, which helps regenerate cellular ATP. Preclinical evidence for creatine's potential neuroprotective effects in animal models of HD has been well-documented. Before the clinical efficacy of creatine can be tested in premanifest HD, its long-term safety and tolerability must be assessed in these individuals and its ability to favorably modify biomarkers of HD should also be confirmed. A two phase protocol is proposed in which 60 premanifest and at-risk subjects will randomized into a double blind placebo controlled dose titration study bringing them to 30 grams daily or their highest tolerated dose. The placebo-controlled phase will permit the detection of toxicity and intolerability due to the active compound (creatine), and enable a dose response assessment of biomarkers. In the second phase, all subjects will enter a year long open-label treatment on 30 grams daily of creatine. This phase will maximize the subjects on active compound to promote recruitment and retention, to expand assessment of safety data on all subjects, and increase the power to detect and measure potential biological markers and any response to the active compound. The clinical impact of creatine will be assessed using the United Huntington's Disease Rating Scale. Safety and tolerability will be assessed by analyzing clinical and laboratory adverse events. Serum levels of creatine will be used to assess compliance and whether there is a relationship between bioavailability and response. 8OH2'dG and related markers will be assessed to determine whether creatine treatment can chronically suppress markers of energy depletion and oxidative injury and whether suppression correlates with slowing the progression of HD. Morphometric MRI will be used to determine whether creatine can slow brain atrophy in premanifest HD. This study will provide the pilot data needed to plan a future study to determine whether creatine can delay the onset or slow the progress of HD in premanifest individuals.

ELIGIBILITY:
Inclusion Criteria:

- Expansion positive or 50% at risk for HD and not diagnosed clinically

Exclusion Criteria:

- Unstable medical conditions

Additional inclusion and exclusion criteria apply.

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Completion of Study (tolerability) | 18 Months
  Tolerability (proportion of subjects completing study at given dose level)
Safety | 18 Months
  Frequency of adverse events

SECONDARY OUTCOMES:
Pharmacokinetic and Pharmacodynamic biomarkers | 18 months
UHDRS | 18 months
Brain Volumetric & Neurochemical Changes | 18 Months
Metabolomics & Gene Expression Biomarkers | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Hersch, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

REFERENCES:
- [Background] Kim J, Amante DJ, Moody JP, Edgerly CK, Bordiuk OL, Smith K, Matson SA, Matson WR, Scherzer CR, Rosas HD, Hersch SM, Ferrante RJ. Reduced creatine kinase as a central and peripheral biomarker in Huntington's disease. Biochim Biophys Acta. 2010 Jul-Aug;1802(7-8):673-81. doi: 10.1016/j.bbadis.2010.05.001. Epub 2010 May 9. PMID 20460152
- [Background] Hersch SM, Gevorkian S, Marder K, Moskowitz C, Feigin A, Cox M, Como P, Zimmerman C, Lin M, Zhang L, Ulug AM, Beal MF, Matson W, Bogdanov M, Ebbel E, Zaleta A, Kaneko Y, Jenkins B, Hevelone N, Zhang H, Yu H, Schoenfeld D, Ferrante R, Rosas HD. Creatine in Huntington disease is safe, tolerable, bioavailable in brain and reduces serum 8OH2'dG. Neurology. 2006 Jan 24;66(2):250-2. doi: 10.1212/01.wnl.0000194318.74946.b6. PMID 16434666
- [Background] Ryu H, Rosas HD, Hersch SM, Ferrante RJ. The therapeutic role of creatine in Huntington's disease. Pharmacol Ther. 2005 Nov;108(2):193-207. doi: 10.1016/j.pharmthera.2005.04.008. Epub 2005 Aug 1. PMID 16055197
- [Background] Dedeoglu A, Kubilus JK, Yang L, Ferrante KL, Hersch SM, Beal MF, Ferrante RJ. Creatine therapy provides neuroprotection after onset of clinical symptoms in Huntington's disease transgenic mice. J Neurochem. 2003 Jun;85(6):1359-67. doi: 10.1046/j.1471-4159.2003.01706.x. PMID 12787055
- [Background] Andreassen OA, Dedeoglu A, Ferrante RJ, Jenkins BG, Ferrante KL, Thomas M, Friedlich A, Browne SE, Schilling G, Borchelt DR, Hersch SM, Ross CA, Beal MF. Creatine increase survival and delays motor symptoms in a transgenic animal model of Huntington's disease. Neurobiol Dis. 2001 Jun;8(3):479-91. doi: 10.1006/nbdi.2001.0406. PMID 11447996
- [Background] Ferrante RJ, Andreassen OA, Jenkins BG, Dedeoglu A, Kuemmerle S, Kubilus JK, Kaddurah-Daouk R, Hersch SM, Beal MF. Neuroprotective effects of creatine in a transgenic mouse model of Huntington's disease. J Neurosci. 2000 Jun 15;20(12):4389-97. doi: 10.1523/JNEUROSCI.20-12-04389.2000. PMID 10844007
- [Background] Stack EC, Dedeoglu A, Smith KM, Cormier K, Kubilus JK, Bogdanov M, Matson WR, Yang L, Jenkins BG, Luthi-Carter R, Kowall NW, Hersch SM, Beal MF, Ferrante RJ. Neuroprotective effects of synaptic modulation in Huntington's disease R6/2 mice. J Neurosci. 2007 Nov 21;27(47):12908-15. doi: 10.1523/JNEUROSCI.4318-07.2007. PMID 18032664
- [Background] Bechtel N, Scahill RI, Rosas HD, Acharya T, van den Bogaard SJ, Jauffret C, Say MJ, Sturrock A, Johnson H, Onorato CE, Salat DH, Durr A, Leavitt BR, Roos RA, Landwehrmeyer GB, Langbehn DR, Stout JC, Tabrizi SJ, Reilmann R. Tapping linked to function and structure in premanifest and symptomatic Huntington disease. Neurology. 2010 Dec 14;75(24):2150-60. doi: 10.1212/WNL.0b013e3182020123. Epub 2010 Nov 10. PMID 21068430
- [Background] Rosas HD, Lee SY, Bender AC, Zaleta AK, Vangel M, Yu P, Fischl B, Pappu V, Onorato C, Cha JH, Salat DH, Hersch SM. Altered white matter microstructure in the corpus callosum in Huntington's disease: implications for cortical "disconnection". Neuroimage. 2010 Feb 15;49(4):2995-3004. doi: 10.1016/j.neuroimage.2009.10.015. Epub 2009 Oct 19. PMID 19850138
- [Background] Rosas HD, Salat DH, Lee SY, Zaleta AK, Hevelone N, Hersch SM. Complexity and heterogeneity: what drives the ever-changing brain in Huntington's disease? Ann N Y Acad Sci. 2008 Dec;1147:196-205. doi: 10.1196/annals.1427.034. PMID 19076442
- [Background] Hersch SM, Rosas HD. Neuroprotection for Huntington's disease: ready, set, slow. Neurotherapeutics. 2008 Apr;5(2):226-36. doi: 10.1016/j.nurt.2008.01.003. PMID 18394565
- [Background] Rosas HD, Salat DH, Lee SY, Zaleta AK, Pappu V, Fischl B, Greve D, Hevelone N, Hersch SM. Cerebral cortex and the clinical expression of Huntington's disease: complexity and heterogeneity. Brain. 2008 Apr;131(Pt 4):1057-68. doi: 10.1093/brain/awn025. Epub 2008 Mar 12. PMID 18337273
- [Background] Rosas HD, Tuch DS, Hevelone ND, Zaleta AK, Vangel M, Hersch SM, Salat DH. Diffusion tensor imaging in presymptomatic and early Huntington's disease: Selective white matter pathology and its relationship to clinical measures. Mov Disord. 2006 Sep;21(9):1317-25. doi: 10.1002/mds.20979. PMID 16755582
- [Background] Rosas HD, Hevelone ND, Zaleta AK, Greve DN, Salat DH, Fischl B. Regional cortical thinning in preclinical Huntington disease and its relationship to cognition. Neurology. 2005 Sep 13;65(5):745-7. doi: 10.1212/01.wnl.0000174432.87383.87. PMID 16157910